CLINICAL TRIAL: NCT01748916
Title: Evaluation of the Effect of the Consumption of Papaya, Tomato, and Carrot on the Bioavailability of Carotenoids
Brief Title: Comparison of Carotenoid Bioavailability From Fresh Papaya, Tomato and Carrot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Hohenheim (Other); Universidad de Costa Rica (Other)
Responsible Party: Principal Investigator, Jessica Cooperstone, Research Scientist, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2011H0336
Record Dates: First submitted 2012-12-03; First posted 2012-12-13 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Focus of Study: Carotenoid Absorption
Keywords: Papaya; Carrot; Tomato; Carotenoids; Lycopene; Beta-carotene; Beta-cryptoxanthin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Papaya-Carrot-Tomato (Experimental): Test meals were consumed in the following order: 1. Papaya 2. Carrot 3. Tomato.
  Interventions: Other: Papaya; Other: Carrot; Other: Tomato
- Papaya-Tomato-Carrot (Experimental): Test meals were consumed in the following order: 1. Papaya 2. Tomato 3. Carrot
  Interventions: Other: Papaya; Other: Carrot; Other: Tomato
- Tomato-Papaya-Carrot (Experimental): Test meals were consumed in the following order: 1. Tomato 2. Papaya 3. Carrot
  Interventions: Other: Papaya; Other: Carrot; Other: Tomato
- Tomato-Carrot-Papaya (Experimental): Test meals were consumed in the following order: 1. Tomato 2. Carrot 3. Papaya
  Interventions: Other: Papaya; Other: Carrot; Other: Tomato
- Carrot-Papaya-Tomato (Experimental): Test meals were consumed in the following order: 1. Carrot 2. Papaya 3. Tomato
  Interventions: Other: Papaya; Other: Carrot; Other: Tomato
- Carrot-Tomato-Papaya (Experimental): Test meals were consumed in the following order: 1. Carrot 2. Tomato 3. Papaya
  Interventions: Other: Papaya; Other: Carrot; Other: Tomato

INTERVENTIONS:
Other: Papaya — Post-prandial study feeding 400-506 g papaya (1.6 mg beta-carotene, 2.1 mg beta-cryptoxanthin, 13 mg lycopene), 150 g yogurt (10% fat), and 45 g of fat free bread.
Other: Carrot — Post-prandial study feeding 25-35 g carrot (= 1.6 mg beta-carotene), 150 g yogurt (10% fat), and 45 g of fat free bread.
Other: Tomato — Post-prandial study feeding 256-396 g tomato (= 13 mg lycopene), 150 g yogurt (10% fat), and 45 g of fat free bread.

SUMMARY:
The goal of this study is to determine if papaya fruits are an exceptionally good food source for carotenoids in humans, particularly when compared more common carotenoid sources like carrots and tomatoes. This objective will be accomplished by quantitation of the immediate post-prandial plasma concentrations of parent carotenoids and vitamin A metabolites from subjects who consumed a meal containing fresh papaya, tomato, and carrot.

DETAILED DESCRIPTION:
The main purpose of this study is comparing bioavailability of papaya carotenoids versus carrot and tomato carotenoids. Previously, vitamin A deposition in rat livers was studied, showing that carotenoid bioavailability from papaya is higher than from spinach, parsley and carrots. Detailed knowledge about human carotenoid absorption and conversion from papaya fruit compared to other food sources is still lacking.

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals

Exclusion Criteria:

* lactating, pregnant, or planned to be pregnant
* smokers/those who use tobacco products
* metabolic or malabsorption disorders
* had a history of cancer
* history of liver insufficiency or other gastro-intestinal diseases
* allergy to papaya, carrots or tomatoes
* obesity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Schwartz, Ph.D., Principal Investigator — Ohio State University
Locations (2):
- The Ohio State University, Columbus, Ohio, United States
- University of Costa Rica, San José, Costa Rica

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was carried out at the University of Costa Rica during June 2011 - August 2011.
Pre-assignment Details: Sixteen healthy, non-pregnant, non-smoking participants (21-44 y) were enrolled after checking eligibility, which was based on a questionnaire. Exclusion criteria included any history of chronic gastrointestinal disease, use of medications affecting lipid metabolism, regular use of carotenoid-containing supplements and frequent alcohol consumption.
Period: Overall Study
Arm/Group | Papaya-Carrot-Tomato | Papaya-Tomato-Carrot | Tomato-Papaya-Carrot | Tomato-Carrot-Papaya | Carrot-Papaya-Tomato | Carrot-Tomato-Papaya
Started | 2 | 3 | 2 | 3 | 3 | 3
Completed | 2 | 3 | 2 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Groups (Average): All study participants
Arm/Group | All Groups (Average)
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 27 [21 to 44]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Region of Enrollment [Number; unit: participants]
  Costa Rica | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of Carotenoid Absorption From Papaya, Carrot and Tomato
Description: The primary goal of this research is to investigate whether papaya can deliver increased quantities of carotenoids when compared to carrot and tomato. An area under the curve for concentration of carotenoids (from triglyceride rich lipoprotein (TRL) fraction of plasma) over time will be determined to quantify absorption, after subjects consume a meal containing papaya, carrot or tomato.
Time Frame: 8 post-prandial blood samples over 9.5 hours
Measure: Median (Inter-Quartile Range); unit: nmol*h/L
Arm/Group | Beta-Carotene Absorption From Papaya | Beta-Carotene Absorption From Tomato | Beta-Carotene Absorption From Carrot | Lycopene Absorption From Papaya | Lycopene Absorption From Tomato
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16
nmol*h/L | 163 [155 to 210] | 62 [28 to 103] | 64 [40 to 96] | 174 [130 to 249] | 58 [47 to 102]

ADVERSE EVENTS:
Groups:
- All Groups: All groups in study
Arm/Group | All Groups
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No